CLINICAL TRIAL: NCT01475292
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Safety and Tolerability of Treatment With Repeat Doses of Inhaled RV568 in Patients With COPD
Brief Title: A Study to Investigate How Safe and Well Tolerated RV568 is in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Respivert Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RVH006; 2011-004031-31 (EudraCT Number)
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- RV568 treatment group low dose (Experimental)
  Interventions: Drug: RV568
- RV568 treatment group high dose (Experimental)
  Interventions: Drug: RV568
- Placebo treatment group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RV568 — RV568 50 ug administered via a nebuliser once daily for 14 days
  Arms: RV568 treatment group low dose
Drug: RV568 — RV568 100 ug administered via a nebuliser once daily for 14 days
  Arms: RV568 treatment group high dose
Drug: Placebo — Placebo administered via a nebuliser once daily for 14 days
  Arms: Placebo treatment group

SUMMARY:
RV568 is being developed as a possible treatment of diseases such as smoking related lung disease (also known as Chronic Obstructive Pulmonary Disease - COPD) and asthma.

The main purpose of this study is to examine the safety of RV568 in COPD patients. Two dose strengths of RV568 and a placebo will be tested in this study, which will be given by inhaling a liquid suspension from a nebuliser once a day for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 40-75 years inclusive at the time of signing the informed consent.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* COPD diagnosis: Subjects with a diagnosis of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines, with symptoms compatible with COPD for at least 1 year prior to screening.
* Severity of Disease: subjects who conform to the current severity classification for GOLD Stage II/III disease in terms of post-bronchodilator spirometry at screening (Post-salbutamol FEV1/FVC ratio of ≤ 0.70 and post-salbutamol FEV1 ≥ 40 % and ≤ 80 % of predicted normal values calculated using ECCS reference equations)
* Demonstrated ability to use the I-neb AAD system at screening.
* Subject is a current or previous smoker with a smoking history of ≥ 10 pack years

Exclusion Criteria:

* A history of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation
* A history of > 1 hospitalisation for COPD in the previous 2 years prior to screening.
* Evidence of cor pulmonale or clinically significant pulmonary hypertension or chronic (in the opinion of the Investigator) use of oxygen.
* Upper or lower respiratory tract infection, including exacerbation of COPD, within 6 weeks of screening.
* Other respiratory disorders: Subjects with a current diagnosis of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases or other active pulmonary diseases.
* Subjects with a history of chronic disease including, but not limited to, sleep apnoea, cardiovascular, endocrine, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, or ophthalmic diseases that the Investigator believes are clinically significant.
* Previous lung resection or lung reduction surgery.
* Pregnant or nursing females.
* Any abnormal or clinically significant ECG or laboratory values that the Investigator considers would put the subject at risk through participation. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included if the Investigator and the sponsor representative agree it is unlikely to introduce additional risk factors and will not interfere with study procedures.
* ALT > 2 x ULN at the screening visit.
* A positive pre-study Hepatitis B surface antigen, positive Hepatitis C antibody result, or positive test for HIV antibody at the screening visit (or within the 3 months prior to screening).
* Positive test for drugs of abuse at screening that cannot be satisfactorily explained by a prescription history (e.g., recent use of codeine tablets).
* History of alcohol abuse within the previous 6 months
* Has had major surgery, (requiring general anesthesia) within 6 weeks before the screening visit, or will not have fully recovered from surgery, or planned surgery through the end of the study
* Participated in any other clinical study of an NCE within 3 months, or in a study of a marketed drug within 1 month (or within 5 half-lives of the NCE or marketed drug, whichever is the longest) of first dose; or has participated in 4 studies in the previous 12 months.
* A disclosed history, or one known to the Investigator, of significant noncompliance in previous investigational studies or with prescribed medications.
* Allergy to any of the active or inactive ingredients in the study medication, or history of drug, or other allergy that, in the opinion of the Investigator or RespiVert medical monitor, would contraindicate their participation.
* Donation of blood in excess of 500 mL within a 3 month period prior to dosing, or if study participation would result in blood loss in excess of 500 mL in a 3 month period.
* Subject is mentally or legally incapacitated.
* Has any condition or are taking a medication that, in the opinion of the Investigator, would make participation not be in the best interest (i.e., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
* Is an employee of the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the Investigator.
* Any other reason that the Investigator considers makes the subject unsuitable to participate.
* Subject has a history of unstable, or uncontrolled hypertension, or has been diagnosed with hypertension in last 6 months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 28 days
  Assessment of vital signs, ECG, adverse event assessment, clinical laboratory screening and spirometry.

SECONDARY OUTCOMES:
Plasma RV568 levels | 0,15,30,45 min and 1,2,4,6,8,10,12 & 24 hours post dose on Days 1 & 14, 0,1 & 2 hours post dose on Day 7 and one time point on Days 4, 21 & 28
Assessment of lung function using a body plethysmograph | 2 week treatment period
Assessment of markers of inflammation in sputum | 2 week treatment period
Assessment of markers of inflammation in blood | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Siew, MD, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital
Locations (2):
- United Kingdom (2):
  - Quintiles Drug Research Unit at Guy's Hospital, London
  - Medicines Evaluation Unit (MEU), Manchester